CLINICAL TRIAL: NCT06038734
Title: Using Point-of-Care-Ultrasound (POCUS) to Assess Gastric Contents Among Fasting Pre-operative Patients Taking GLP-1 Agonists.
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 23-0578
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-09

CONDITIONS: Delayed Gastric Emptying; Gastroparesis
Keywords: GLP-1 agonists; retained gastric contents; glucagon-like peptide receptor-1 agonists; perioperative
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GLP-1 agonists: Pre-operative gastric ultrasound to evaluate for retained gastric contents in appropriately fasted patients who are using GLP-1 agonist medications.
  Interventions: Diagnostic Test: gastric ultrasound
- Control: Pre-operative gastric ultrasound to evaluate for retained gastric contents in appropriately fasted patients who are not using GLP-1 agonist medications.
  Interventions: Diagnostic Test: gastric ultrasound

INTERVENTIONS:
Diagnostic Test: gastric ultrasound — Utilize POC gastric ultrasound to identify the presence of retained gastric contents.

SUMMARY:
Given the increased prescription of GLP-1 agonists for both diabetes and obesity management and the implications of the proposed delayed gastric emptying in the setting of an anesthetic, it is critical to determine if patients taking GLP-1 agonists have an increased rate of delayed gastric emptying. The purpose of this prospective gastric ultrasound evaluation of pre-operative patients is to determine the incidence of a full stomach despite a standard pre-operative fasting period.

ELIGIBILITY:
Inclusion Criteria:

* GLP-1 agonist use within previous 30 days
* Appropriately fasted per standard guidelines

Exclusion Criteria:

* History of gastric surgery / gastric volume reduction
* Critical illness
* Inability to provide informed consent
* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include non-critically ill adults 18 years and older undergoing various elective surgical procedures at the University of North Carolina Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Retained gastric contents | At time of pre-operative assessment
  Presence of retained gastric contents, either liquid or solid

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Gouker, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Medical Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.